CLINICAL TRIAL: NCT05159440
Title: A Phase 1, First in Human, Dose-Escalation Study of TORL-2-307-MAB in Participants With Advanced Cancer
Brief Title: First in Human Study of TORL-2-307-MAB in Participants With Advanced Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TORL Biotherapeutics, LLC (Industry)
Collaborators: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TORL2307MAB-001
Record Dates: First submitted 2021-12-01; First posted 2021-12-16 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor; Gastric Cancer; Pancreas Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: claudin18.2
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy Dose Dose Finding - Part 1 (Experimental): TORL-2-307-MAB
  Interventions: Drug: TORL-2-307-MAB
- Expansion as Monotherapy - Part 2 (Experimental): TORL-2-307-MAB
  Interventions: Drug: TORL-2-307-MAB

INTERVENTIONS:
Drug: TORL-2-307-MAB — monoclonal antibody

SUMMARY:
This first-in-human study will evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of TORL-2-307-MAB in patients with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor
* Measurable disease, per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function

Exclusion Criteria:

* Has not recovered [recovery is defined as NCI CTCAE, version 5.0, grade ≤1] from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements
* Received prior chemotherapeutic, investigational, or other therapies for the treatment of cancer within 14 days with small molecule and within 28 days with biologic before the first dose of TORL-2-307-MAB
* Progressive or symptomatic brain metastases
* Serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection
* History of significant cardiac disease
* History of myelodysplastic syndrome (MDS) or AML
* History of another cancer within 3 years before Day 1 of study treatment, with the exception of basal or squamous cell carcinoma of the skin that has been definitively treated. A history of other malignancies with a low risk of recurrence, including appropriately treated ductal carcinoma in situ (DCIS) of the breast and prostate cancer with a Gleason score less than or equal to 6, are also not excluded
* If female, is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events | up to 2 years
  Incidence and severity of adverse events, serious adverse events, according to NCI-CTCAE Version 5.0
Maximum Tolerated Dose (MTD) | 28 Days
  Highest administered dose with < 33% participants experiencing dose limiting toxicity (DLT) in the first 6 DLT evaluable participants
Recommended Phase 2 Dose (RP2D) | up to 2 years
  Based on the maximum tolerated dose, cumulative safety, and pharmacokinetic data

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 2 years
  Percentage of participants with best response of complete response (CR) or partial response (PR) according to RECIST 1.1
Duration of Response (DOR) | up to 2 years
  Time from CR or PR to objective disease progression or death to any cause
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time from the start of the treatment until objective disease progression or death from any cause
Time to Response (TTR) | up to 2 years
  Time from start of treatment to complete response or partial response
1 Year Overall Survival (1YOS) | 1 year
  Proportion of participants alive at 1 year from the start of treatment to death from any cause
2 Year Overall Survival (2YOS) | 2 years
  Proportion of participants alive at 2 years from the start of treatment to death from any cause
Number of anti-drug antibody (ADA) Positive Participants | up to 2 years
  Immunogenicity will be measured by the number of participants that are ADA positive.
Maximum Serum Concentration of TORL-2-307-MAB (Cmax) | 21 days
  PK assessment
Minimum Serum Concentration of TORL-2-307-MAB (Cmin) | 21 days
  PK assessment
Maximum Serum Concentration of TORL-2-307-MAB at Steady State (Cmax,ss) | 63 days
  PK assessment
Minimum Serum Concentration of TORL-2-307-MAB at Steady State (Cmin,ss) | 63 days
  PK assessment
Time of Maximum Serum Concentration of TORL-2-307-MAB (Tmax) | 21 days
  PK assessment
Time of Minimum Serum Concentration of TORL-2-307-MAB (Tmin) | 21 days
  PK Assessment
Time of Minimum Serum Concentration of TORL-2-307-MAB at Steady State (Tmin,ss) | 63 days
  PK Assessment
Terminal Half-life (t1/2) of Serum TORL-2-307-MAB | 63 days
  PK Assessment
Area under the Serum Concentration-Time curve from the time of dosing to the last measurable concentration (AUClast) for TORL-2-307-MAB | 21 days
  PK Assessment
Area under the Serum Concentration-Time curve from the time of dosing extrapolated to time infinity (AUCinf) for TORL-2-307-MAB | 63 days
  PK Assessment
Apparent volume of distribution during the terminal phase (Vz) of TORL-2-307-MAB | 63 days
  PK Assessment
Clearance (CL) of TORL-2-307-MAB | 63 days
  PK Assessment
Accumulation ratio (Rac) of TORL-2-307-MAB | 63 days
  PK Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Letrent, PharmD, PhD, Study Director — TORL Biotherapeutics, LLC
Locations (8):
- United States (5):
  - Providence St. Jude Medical Center, Fullerton, California
  - UCLA - JCCC Clinical Research Unit, Los Angeles, California
  - Torrance Memorial Medical, Torrance, California
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Washington University School of Medicine-Siteman Cancer Center, St Louis, Missouri
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul National University Bundang Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Brien NA, McDermott MSJ, Zhang J, Gong KW, Lu M, Hoffstrom B, Luo T, Ayala R, Chau K, Liang M, Madrid AM, Donahue TR, Glaspy JA, Presta L, Slamon DJ. Development of a Novel CLDN18.2-directed Monoclonal Antibody and Antibody-Drug Conjugate for Treatment of CLDN18.2-Positive Cancers. Mol Cancer Ther. 2023 Dec 1;22(12):1365-1375. doi: 10.1158/1535-7163.MCT-23-0353. PMID 37788341